CLINICAL TRIAL: NCT00936741
Title: An Open Label Extension Study of the Efficacy and Safety of CORLUX® (Mifepristone) in the Treatment of the Signs and Symptoms of Endogenous Cushing's Syndrome
Brief Title: An Extension Study of CORLUX in the Treatment of Endogenous Cushing's Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-1073-415
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-02

CONDITIONS: Cushing's Syndrome
Keywords: Cushing's Disease; Cushing's Syndrome; Cushings; Pituitary; ACTH; Adrenocorticotropic hormone; Ectopic; Adrenal adenoma; Adrenal carcinoma; Adrenal autonomy; Cortisol; Hypercortisolemia; Cushingoid; Moon facies; Dorsocervical fat; Plethora; Hirsutism; Violaceous striae; Hormone; Contraceptive; Endocrine; Cushing Syndrome; Ectopic ACTH Secretion
MeSH Terms: conditions — Cushing Syndrome; Pituitary ACTH Hypersecretion; Pituitary Diseases; Choristoma; ACTH Syndrome, Ectopic; Adrenal Cortex Neoplasms; Hirsutism | interventions — Mifepristone; Corlux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mifepristone (Experimental): Mifepristone 300mg to 1200mg once daily
  Interventions: Drug: mifepristone

INTERVENTIONS:
Drug: mifepristone — Mifepristone 300 mg to 1200 mg once daily
  Other Names: CORLUX

SUMMARY:
Participants in study C-1073-400 (NCT00569582) will be invited to participate in this extension study to examine the long term safety of mifepristone in the treatment of the signs and symptoms of endogenous Cushing's syndrome. Total treatment duration may be up to 12 months or longer at the discretion of the Investigator.

DETAILED DESCRIPTION:
Up to 50 subjects will receive mifepristone daily. Subjects completing 24 weeks of mifepristone treatment under Corcept protocol C1073-400 (NCT00569582) will be eligible to continue treatment for an additional 1 year. Assessments of safety, as evaluated by physical examinations, vital signs, laboratory tests and adverse events, will be made. Persistence of improvement in response to mifepristone treatment will also be evaluated during this extension study by assessing the continued or sustained improvement in the signs and symptoms of Cushing's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the Week 24 visit and the 6-Week Follow-up visit of Corcept Study C-1073-400 (NCT00569582).
* In the opinion of the Investigator, are expected to maintain clinical benefit from mifepristone.
* Women of childbearing potential have a negative serum pregnancy test at Entry.
* Women of childbearing potential must be willing to use non-hormonal, medically acceptable methods of contraception during the study.
* Are able to provide written informed consent
* Are able to return to the investigative site to complete the study evaluations outlined in the protocol.
* Will not use systemic estrogens during the study.

Exclusion Criteria:

* Have an acute or unstable medical problem, which could be aggravated by mifepristone treatment.
* Are taking medications within 14 days of the Entry visit that a) have a large first pass metabolism that is largely mediated by CYP3A4 and which have a narrow therapeutic margin; and/or b) are strong CYP3A4 inhibitors.
* Female patients of reproductive potential, who are pregnant or who are unable or unwilling to use medically acceptable, non-hormonal methods of contraception during the study.
* Have received investigational treatment (drug, biological agent or device) other than CORLUX (mifepristone) within 30 days of Entry
* Have a history of an allergic reaction or intolerance to CORLUX (mifepristone)
* Have uncorrected hypokalemia (potassium level of <3.5 mEq/L) at Entry. Spironolactone or eplerenone is allowed to control hypokalemia.
* Postmenopausal women with a history of endometrial hyperplasia with atypia or pathological features consistent with endometrial carcinoma.
* Thickened endometrium on the Entry Visit transvaginal ultrasound that has not resolved after induction of menstrual bleeding with progesterone.
* Uncontrolled, clinically significant hypothyroidism or hyperthyroidism.
* Any woman with an intact uterus who has a hemorrhagic disorder or is being treated with an anticoagulant (e.g. warfarin, heparin).
* Have renal failure as defined by a serum creatinine of ≥2.2 mg/dL.
* Elevated total bilirubin >1.5 ULN, elevated ALT or AST ≥3X the upper limit of normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Coleman Gross, MD, Study Director — Corcept Therapeutics
Locations (15):
- United States (15):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - AMCR Institute Inc., Escondido, California
  - Stanford University Medical Center, Stanford, California
  - The Center for Diabetes and Endocrine Care, Hollywood, Florida
  - Northwestern University Feinberg Medical; Division of Endocrinology, Metabolism & Molecular Medicine, Chicago, Illinois
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of New Mexico, Albuquerque, New Mexico
  - Cleveland Clinic Foundation; Dept of Endocrinology, Diabetes & Metabolism, Cleveland, Ohio
  - Oklahoma Diabetes Center, Oklahoma City, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Endocrinology Center at Community Medical Commons, Menomonee Falls, Wisconsin

REFERENCES:
- [Derived] Fein HG, Vaughan TB 3rd, Kushner H, Cram D, Nguyen D. Sustained weight loss in patients treated with mifepristone for Cushing's syndrome: a follow-up analysis of the SEISMIC study and long-term extension. BMC Endocr Disord. 2015 Oct 27;15:63. doi: 10.1186/s12902-015-0059-5. PMID 26507877
- [Derived] Fleseriu M, Findling JW, Koch CA, Schlaffer SM, Buchfelder M, Gross C. Changes in plasma ACTH levels and corticotroph tumor size in patients with Cushing's disease during long-term treatment with the glucocorticoid receptor antagonist mifepristone. J Clin Endocrinol Metab. 2014 Oct;99(10):3718-27. doi: 10.1210/jc.2014-1843. Epub 2014 Jul 11. PMID 25013998
- See also: Corcept C-1073-400 Clinicaltrials.gov Study Listing — http://clinicaltrials.gov/ct2/show/NCT00569582

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects completing 24 weeks of mifepristone treatment under Corcept protocol C1073-400 (NCT00569582) were eligible to continue treatment in C1073-415 at the dose being administered at the end of treatment in C1073-400 (NCT00569582).
Pre-assignment Details: Only subjects who had completed C1073-400 (NCT00569582) were enrolled. All subjects received active drug (no placebo).
Groups:
- Open-label: mifepristone at doses from 300 mg/day up to 1200 mg/day daily
Period: Overall Study
Arm/Group | Open-label
Started | 30
Completed | 21
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Open-label
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Subjects who received at least one dose of mifepristone were included in the safety analysis.
Time Frame: Up to three years.
Population: Subjects who received one dose of study drug were included in the safety and ITT analyses.
Measure: Number; unit: participants
Arm/Group | Open-label
Number analyzed (Participants) | 30
participants | 30

2. Secondary Outcome: The Long-term Benefit of Mifepristone Treatment in Cushing's Syndrome as Measured by Changes in the Score on the Physician's Global Assessment of Disease Severity
Description: The mean Investigator's rating of the change in subject's signs and symptoms of Cushing's syndrome from Baseline (Entry into C1073-415) to Endpoint on the Physician's Global Assessment of Disease Severity was ranked on a 9-point scale (9 = much worse, 7 = worse, 5 = no change, 3 = better, 1 = much better). Higher scores indicate more severe illness. Scoring was done at all visits except the 6 Week Follow-up visit; the final visit result (Endpoint) is reported here.
  The instruction was "Rate the change in the subject's signs and symptoms of Cushing's from Baseline (1 = much better to 9 = much worse)".
Time Frame: Up to three years.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label
Number analyzed (Participants) | 30
units on a scale | 3.3 (1.74)

ADVERSE EVENTS:
Time Frame: up to 36 months from entry.
Groups:
- Mifepristone 300 to 1200 mg Daily: mifepristone at doses from 300 mg/day to 1200 mg/day
Arm/Group | Mifepristone 300 to 1200 mg Daily
Serious Adverse Events (participants affected / at risk) | 18/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone 300 to 1200 mg Daily (N=30)
Pericarditis (Cardiac disorders) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Amyloidosis (Immune system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Arthritis Bacterial (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood Postassium Decreased (Investigations) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone 300 to 1200 mg Daily (N=30)
Adrenal insufficiency (Endocrine disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 15 (29)
Vomiting (Gastrointestinal disorders) | 7 (14)
Fatique (General disorders) | 12 (14)
Oedema peripheral (General disorders) | 7 (10)
Nasopharyngitis (Infections and infestations) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 6 (7)
Blood potassium decreased (Investigations) | 14 (46)
Thyroid function test abnormal (Investigations) | 6 (6)
Headache (Nervous system disorders) | 11 (22)
Dizziness (Nervous system disorders) | 7 (9)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 4 (6)
Tachycadia (Cardiac disorders) | 3 (3)
Cushing's syndrome (Endocrine disorders) | 2 (2)
Gynaecomastia (Endocrine disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 3 (3)
Cataract nuclear (Eye disorders) | 2 (3)
Diplopia (Eye disorders) | 2 (2)
Vision blurred (Eye disorders) | 2 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Toothache (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 2 (4)
Pneumonia (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (7)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)
Androgens increased (Investigations) | 2 (3)
Blood cholesterol increased (Investigations) | 4 (4)
Blood corticotrophin increased (Investigations) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2)
Blood potassium increased (Investigations) | 2 (3)
Blood testosterone free increased (Investigations) | 3 (4)
Blood testosterone increased (Investigations) | 3 (3)
Electrocardiogram QT prolonged (Investigations) | 3 (3)
Protein urine (Investigations) | 2 (2)
Urine cortisol / creatinine ratio increased (Investigations) | 2 (3)
White blood cell count increased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (4)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pituitary tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Muscular weakness (Nervous system disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 3 (5)
Insomnia (Psychiatric disorders) | 4 (4)
Panic attack (Psychiatric disorders) | 2 (2)
Sleep disorder (Psychiatric disorders) | 2 (3)
Nephrolithiasis (Renal and urinary disorders) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 2 (2)
Endometrial disorder (Reproductive system and breast disorders) | 4 (7)
Endometrial hypertrophy (Reproductive system and breast disorders) | 10 (12)
Metrorrhagia (Reproductive system and breast disorders) | 4 (5)
Ovarian cyst (Reproductive system and breast disorders) | 2 (4)
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 (2)
Hot flush (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 9 (14)
Hypotension (Vascular disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days